CLINICAL TRIAL: NCT01435018
Title: A Randomized Comparison of Three Regimens of Chemotherapy With Compatible Antiretroviral Therapy for Treatment of Advanced AIDS-KS in Resource-Limited Settings
Brief Title: Three Chemo Regimens as an Adjunct to ART for Treatment of Advanced AIDS-KS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Cancer Institute (NCI) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH); AIDS Malignancy Consortium (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5263/AMC 066; 1U01AI068636 (NIH); U01CA121947 (NIH)
Record Dates: First submitted 2011-09-14; First posted 2011-09-15 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-09

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Etoposide; Bleomycin; Vincristine; Paclitaxel; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ET+ART (Experimental): Etoposide (ET) plus co-formulated Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate (EFV/FTC/TDF)
  Interventions: Drug: Etoposide (ET); Drug: Co-formulated Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate (EFV/FTC/TDF)
- BV+ART (Experimental): Bleomycin and Vincristine (BV) plus co-formulated Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate (EFV/FTC/TDF)
  Interventions: Drug: Bleomycin and Vincristine (BV); Drug: Co-formulated Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate (EFV/FTC/TDF)
- PTX+ART (Active Comparator): Paclitaxel (PTX) plus co-formulated Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate (EFV/FTC/TDF)
  Interventions: Drug: Paclitaxel (PTX); Drug: Co-formulated Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate (EFV/FTC/TDF)

INTERVENTIONS:
Drug: Etoposide (ET) — Beginning on day one of the chemotherapy cycle, ET was given orally in a dose of 50 mg twice daily for 7 consecutive days for the first cycle. If there was no Grade >= 2 toxicity attributable to ET after the first cycle, the dose was escalated to 150 mg daily for 7 days in divided doses of 100 mg/50 mg for the second cycle. After the second cycle, if there was no Grade >= 2 toxicity attributable to ET, the dose was escalated to 100 mg twice daily for 7 days for the third and subsequent cycles.
  Treatment with ET was continued for six cycles at the maximum dose achieved or until toxicity requiring discontinuation of study chemotherapy, or the site investigator, after consulting with the protocol CMC, had determined that alternative therapy is required, whichever occurs first.
  Arms: ET+ART
Drug: Bleomycin and Vincristine (BV) — BV was administered on day one of each chemotherapy cycle.
  Vincristine sulfate was administered at a dose of 2 mg (fixed dose) in a volume of 2 mL over 1 minute into the sidearm of a rapidly flowing intravenous infusion every 3 weeks. The vincristine infusion was followed by bleomycin as detailed below.
  Bleomycin sulfate was administered at a dose of 15 units/m^2 over 10 minutes every 3 weeks.
  Treatment with BV was continued for six cycles, or until toxicity requiring discontinuation of study chemotherapy, or the site investigator, after consulting with the protocol CMC, had determined that alternative therapy is required, whichever occurs first.
  Arms: BV+ART
Drug: Paclitaxel (PTX) — Paclitaxel was administered by IV infusion in 200 mL, 250 mL, or 500 mL of 5% dextrose or 0.9%Sodium Chloride for injection at a dose of 100 mg/m^2 body surface area (BSA) every 3 weeks.
  Arms: PTX+ART
Drug: Co-formulated Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate (EFV/FTC/TDF) — The following ART regimens were used:
  1. EFV/FTC/TDF (Atripla) 200 mg/300 mg/600 mg orally once daily at bedtime or
  2. FTC/TDF 200 mg/300 mg (Truvada) orally once daily at bedtime plus EFV (Stocrin) 600 mg orally once daily at bedtime or
  3. FTC/TDF 200 mg/300 mg (Truvada) orally once daily plus nevirapine (NVP) 200 mg orally twice daily or
  4. FTC/TDF 200 mg/300 mg (Truvada) orally once daily plus PI/r at standard dosing or
  5. FTC/TDF 200 mg/300 mg (Truvada) orally once daily plus integrase inhibitor at standard dosing

SUMMARY:
This study was done to compare the safety and efficacy of three combination treatments for Kaposi's Sarcoma (KS) and AIDS:

1. Etoposide (ET) plus co-formulated Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate (EFV/FTC/TDF) (ET+ART),
2. Bleomycin and Vincristine (BV) plus co-formulated EFV/FTC/TDF (BV+ART),
3. Paclitaxel (PTX) plus co-formulated EFV/FTC/TDF (PTX+ART).

DETAILED DESCRIPTION:
The study consisted of four steps. Study duration was up to 240 weeks.

At the study Step 1 entry, participants were randomized with equal probability to each of the three regimens (ET+ART, BV+ART, PTX+ART). The original target sample size was 706. Randomization was stratified by:

1. Screening CD4 lymphocyte cell count (<100, >=100 cells/mm³), and
2. Country.

For participants who had an initial Independent Endpoint Review Committee (IERC) confirmed KS response and subsequent IERC-confirmed KS progression, and who, in the opinion of the investigator and with concurrence of the protocol Clinical Management Committee (CMC), could potentially have benefitted from another course of the same chemotherapy utilized in Step 1, entered Step 2. (Please see details on Step 2 eligibility.)

In Step 3, participants were randomized with equal probability to one of the two chemotherapy arms not utilized in Step 1. (Please see details on Step 3 eligibility.)

In Step 4, participants were assigned to the remaining study-provided chemotherapy not given in Step 1, Step 2 or Step 3. (Please see details on Step 4 eligibility.)

Step 1 visits occurred at screening, entry and weeks 3, 6, 9, 12, 15, 18, 21,24, 27, 30, 33, 36, 39, 42, 45, 48, 60, 72, 84 and 96 from study entry. Visits for Steps 2, 3 and 4 were scheduled at entry and weeks 3, 6, 9, 12, 15, 18, 21,24, 27, 30, 33, 36, 39, 42, 45, 48, 60, 72, 84 and 96 from the corresponding step entry date. Key evaluations included targeted physical examination, clinical assessment, KS examination, hematology, chemistry, pregnancy testing (for women of reproductive potential), and pulse oximetry for participants on BV+ART. CD4 count and HIV viral load were obtained every 12 weeks. Assessment of peripheral neuropathy was done at screening, weeks 9 and 21, and for those on BV+ART or PTX+ART, additionally at weeks 3, 6, 15 and 18. KS tumor punch biopsy, serum, plasma and peripheral blood mononuclear cells (PBMCs) were obtained and stored for use in future analyses. Participants also completed ET and ART adherence evaluations and quality of life questionnaires.

Enrollment to ET+ART and initiation of ET+ART in subsequent steps were discontinued in March 2016, based on the recommendation of the Data and Safety Monitoring Board (DSMB) due to ET+ART being less effective than PTX+ART. No safety concerns were identified. ET+ART participants in Step 1 or Step 2, in discussion with the local investigator and in consultation with the protocol CMC, could discontinue ET and enter Step 3. ET+ART participants in Step 3 could discontinue ET and start the remaining chemotherapy regimen in Step 4 in discussion with the local investigator and in consultation with the protocol CMC. Unless otherwise indicated, comparison between ET+ART and PTX+ART was based on the March 2016 data. The study remained open to enrollment and the remaining participants were randomized at Step 1 entry between BV+ART and PTX+ART. The target total sample size was revised to 446.

The DSMB recommended stopping the study in March 2018 due to BV+ART being inferior to PTX+ART. No safety concerns were identified. Study accrual was stopped. Eligible Step 1 PTX+ART participants entered Step 2 to receive PTX+ART; Step 1 and Step 2 BV+ART participants eligible to receive PTX+ART moved to Step 3 to receive PTX+ART. Otherwise, participants permanently transitioned to local care upon arrangement of appropriate oncology and ART, and then went off study. Participants who received ET while on study were followed for 144 weeks after beginning the last cycle of ET.

Comparison between BV+ART and PTX+ART was based on the March 2018 data.

ELIGIBILITY:
Inclusion Criteria for Step 1:

1. HIV-1 infection
2. Biopsy diagnostic of KS at any time prior to study entry.
3. Current KS stage T1 using ACTG criteria.
4. A minimum of five indicator KS cutaneous marker lesions (or if fewer than five marker lesions are available, the total surface area of the marker lesion(s) must be >=700 mm^2) plus an additional two lesions greater or equal to 4x4 mm that are accessible for punch biopsy.
5. CD4+ lymphocyte cell count obtained within 28 days prior to study entry at a DAIDS-approved laboratory.
6. Certain laboratory values, as defined in the protocol, obtained within 14 days prior to study entry.
7. Female study volunteers of reproductive potential must have a negative serum or urine pregnancy test with a sensitivity of 15-25 mIU/mL performed within 48 hours before initiating the protocol-specified medications.
8. All participants must agree not to participate in a conception process (active attempt to become pregnant or to impregnate, donate sperm, in vitro fertilization).
9. If participating in sexual activity that could lead to pregnancy, participant must agree that two reliable forms of contraceptives will be used simultaneously while receiving protocol-specified medications, and for 12 weeks after stopping the medications. Study volunteers who are not of reproductive potential (women who have been post-menopausal for at least 24 consecutive months or have undergone hysterectomy and/or bilateral oophorectomy or men who have documented azoospermia) are eligible without requiring the use of contraceptives.
10. Ability to swallow oral medications and adequate venous access.
11. Karnofsky performance status >= 60 within 28 days prior to entry.
12. Ability and willingness of participant or legal guardian/representative to provide informed consent.

Exclusion Criteria for Step 1:

1. Current chronic, acute, or recurrent serious infections for which the participant has not completed at least 14 days of therapy prior to study entry and/or is not clinically stable.
2. Serious illness requiring systemic treatment and/or hospitalization within 14 days prior to entry.
3. Current or history of known pulmonary fibrosis, chronic obstructive pulmonary disease (COPD), emphysema, bronchiectasis, or diffuse or significant local radiographic interstitial infiltrates on chest x-ray (CXR) or computed axial tomography (CT) scan.
4. Oxygen saturation less than 90% and/or exercise desaturation greater than 4% within 14 days prior to study enrollment.
5. Grade >=3 peripheral neuropathy (PN) at entry.
6. Breastfeeding.
7. Receipt of ART for more than 42 days immediately prior to entry.
8. Prior or current systemic or locally administered chemotherapy.
9. Prior or current radiation therapy.
10. Prior or current immunotherapy, e.g., interferon alfa.
11. Corticosteroid use at doses above those given as replacement therapy for adrenal insufficiency within the last 30 days prior to study entry.
12. Any immunomodulator, HIV vaccine, live attenuated vaccines, or other investigational therapy or investigational vaccine within 30 days prior to study entry.
13. Known allergy/sensitivity or any hypersensitivity to components of study drugs or their formulation.
14. Active drug or alcohol use or dependence that would interfere with adherence to study requirements.
15. Current or anticipated receipt of any of the prohibited medications listed in section 5.5.2 of the protocol.
16. In the opinion of the investigator, any psychological or social condition, or addictive disorder that would preclude compliance with the protocol.

Inclusion Criteria for Step 2:

1. IERC-confirmed complete response (CR) or partial response (PR) to the chemotherapy regimen used in Step 1.
2. IERC-confirmed KS progression at least 12 weeks after the last dose of Step 1 chemotherapy.
3. Fewer than 72 weeks after Step 1 entry
4. Certain laboratory values, as defined in the protocol, obtained within 14 days prior to Step 2 entry.
5. For females of reproductive potential or females not of reproductive potential who do not have required documentation, negative serum or urine pregnancy test with a sensitivity of 15-25 mIU/mL within 7 days prior to Step 2 entry.
6. Karnofsky performance status >=50 within 28 days prior to Step 2
7. All participants must agree not to participate in a conception process (active attempt to become pregnant or to impregnate, donate sperm, in vitro fertilization).

Exclusion Criteria Step 2:

1. Current chronic, acute, or recurrent infections that are serious, in the opinion of the site investigator, for which the participant has not completed at least 14 days of therapy prior to Step 2 entry and/or is not clinically stable.
2. Severe toxicity to the chemotherapy regimen used in Step 1 requiring discontinuation of study chemotherapy.
3. Serious illness, other than progressive KS, requiring systemic treatment and/or hospitalization within 14 days prior to Step 2 entry.
4. For volunteers who received bleomycin in Step 1

   * Development of of pulmonary fibrosis, COPD, emphysema, bronchiectasis, and diffuse or significant local radiographic interstitial infiltrates on CXR or CT scan that in the opinion of the site investigator would exclude bleomycin use.
   * Oxygen saturation less than 90% or exercise desaturation greater than 4% within the last 30 days prior to Step 2 entry.
5. For volunteers who received Vincristine or Paclitaxel in Step 1, Grade >=3 PN at Step 2 entry.
6. Breastfeeding.
7. Other concurrent chemotherapy, immunotherapy, or radiotherapy.
8. Systemic corticosteroid use at doses above those given as replacement therapy for adrenal insufficiency within 30 days of Step 2 entry.
9. Receipt of Etoposide (ET) in Step 1.

Inclusion Criteria Step 3:

1. (a) IERC-confirmed KS progression at any time during Step 1 chemotherapy, or (b) IERC-confirmed KS progression fewer than 12 weeks after the last chemotherapy dose in Step 1 in participants who have had an IERC-confirmed CR or PR, or (c) IERC-confirmed KS progression following Step 1 chemotherapy, without any prior response, or (d) IERC-confirmed KS progression in Step 2, or (d) with concurrence of the CMC, there is dose-limiting toxicity after receiving fewer than four cycles of chemotherapy in Step 1 or Step 2, in the absence of a CR or PR, or (e) volunteers otherwise eligible for Step 2 who, in the opinion of the investigator and with concurrence of the CMC, are unlikely to benefit from another course of the same chemotherapy received in Step 1.
2. Fewer than 72 weeks after Step 1 entry.
3. Certain laboratory values, as defined in the protocol, obtained within 14 days prior to Step 3 entry.
4. For females of reproductive potential or females not of reproductive potential who do not have required documentation, negative serum or urine pregnancy test with a sensitivity of 15-25 mIU/mL within 7 days prior to Step 3 entry.
5. Karnofsky performance status >=50 within 28 days prior to Step 3 entry.
6. All participants must agree not to participate in a conception process (active attempt to become pregnant or to impregnate, donate sperm, in vitro fertilization).

Exclusion Criteria Step 3:

1. Current chronic, acute, or recurrent infections that are serious, in the opinion of the site investigator, for which the participant has not completed at least 14 days of therapy prior to Step 3 entry and/or is not clinically stable.
2. Serious illness, other than progressive KS, requiring systemic treatment and/or hospitalization within 14 days prior to Step 3 entry.
3. Eligible for Step 2 entry.
4. For participants who did not receive bleomycin in Step 1 or Step 2:

   * Development of pulmonary fibrosis, COPD, emphysema, bronchiectasis, and diffuse or significant local radiographic interstitial infiltrates on CXR or CT scan that in the opinion of the site investigator would exclude bleomycin use.
   * Oxygen saturation less than 90% or exercise desaturation greater than 4% within the last 30 days prior to Step 3 entry.
5. Grade >=3 PN at Step 3 entry.
6. Breastfeeding
7. Other concurrent chemotherapy, immunotherapy, or radiotherapy.
8. Systemic corticosteroid use at doses above those given as replacement therapy for adrenal insufficiency within 30 days of Step 3 entry.

Inclusion Criteria Step 4:

1. (a) IERC-confirmed KS progression in Step 3, or (b) With concurrence of the CMC, dose-limiting toxicity after receiving fewer than four cycles of chemotherapy in Step 3, in the absence of a CR or PR, or (c) Current receipt of ET in Step 3.
2. Fewer than 72 weeks after Step 1 entry.
3. Certain laboratory values, as defined in the protocol, obtained within 14 days prior to Step 4 entry.
4. For females of reproductive potential or females not of reproductive potential who do not have required documentation, negative serum or urine pregnancy test with a sensitivity of 15-25 mIU/mL within 7 days prior to Step 4 entry.
5. Karnofsky performance status >=50 within 28 days prior to Step 4 entry.
6. All participants must agree not to participate in a conception process (active attempt to become pregnant or to impregnate, donate sperm, in vitro fertilization).
7. Receipt of ET in Step 1, Step 2, or Step 3.

Exclusion Criteria Step 4:

1. Current chronic, acute, or recurrent infections that are serious, in the opinion of the site investigator, for which the participant has not completed at least 14 days of therapy prior to Step 4 entry and/or is not clinically stable.
2. Serious illness, other than progressive KS, requiring systemic treatment and/or hospitalization within 14 days prior to Step 4 entry.
3. For participants who did not receive bleomycin in Step 1, Step 2, or Step 3:

   * Development of pulmonary fibrosis, COPD, emphysema, bronchiectasis, and diffuse or significant local radiographic interstitial infiltrates on CXR or CT scan that in the opinion of the site investigator would exclude bleomycin use.
   * Oxygen saturation less than 90% or exercise desaturation greater than 4% within the last 30 days prior to Step 4 entry.
4. Grade >=3 PN at Step 4 entry.
5. Breastfeeding.
6. Other concurrent chemotherapy, immunotherapy, or radiotherapy.
7. Systemic corticosteroid use at doses above those given as replacement therapy for adrenal insufficiency within 30 days of Step 4 entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2019-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Borok-Williams, MD, Study Chair — University of Zimbabwe; Susan E. Krown, MD, Study Chair — AIDS Malignancy Consortium
Locations (11):
- Instituto de Pesquisa Clinica Evandro Chagas (12101), Rio de Janeiro, Brazil
- Kenya (3):
  - Moi University International Clnical Trials Unit, Eldoret
  - KMRI / Walter Reed Project Clinical Research Center, Kericho
  - Kenya Medical Research Institute/Center for Disease Control (KEMRI/CDC) CRS (31460), Kisumu
- Malawi (2):
  - Univ. of Malawi, John Hopkins Project, Blantyre
  - Malawi CRS (12001), Lilongwe
- South Africa (3):
  - Family Clinical Research Unit (FAM-CUR) CRS (8950), Cape Town, West Cape
  - Durban Adult HIV CRS (11201), Durban
  - University of Witwatersrand, Johannesburg
- Uganda Cancer Institute ACTG CRS, Kampala, Uganda
- UZ-Parirenyatwa CRS (30313), Harare, Zimbabwe

REFERENCES:
- [Background] Krown SE, Metroka C, Wernz JC. Kaposi's sarcoma in the acquired immune deficiency syndrome: a proposal for uniform evaluation, response, and staging criteria. AIDS Clinical Trials Group Oncology Committee. J Clin Oncol. 1989 Sep;7(9):1201-7. doi: 10.1200/JCO.1989.7.9.1201. PMID 2671281
- [Background] Cianfrocca M, Cooley TP, Lee JY, Rudek MA, Scadden DT, Ratner L, Pluda JM, Figg WD, Krown SE, Dezube BJ. Matrix metalloproteinase inhibitor COL-3 in the treatment of AIDS-related Kaposi's sarcoma: a phase I AIDS malignancy consortium study. J Clin Oncol. 2002 Jan 1;20(1):153-9. doi: 10.1200/JCO.2002.20.1.153. PMID 11773164
- [Result] Krown SE, Moser CB, MacPhail P, Matining RM, Godfrey C, Caruso SR, Hosseinipour MC, Samaneka W, Nyirenda M, Busakhala NW, Okuku FM, Kosgei J, Hoagland B, Mwelase N, Oliver VO, Burger H, Mngqibisa R, Nokta M, Campbell TB, Borok MZ; A5263/AMC066 protocol team. Treatment of advanced AIDS-associated Kaposi sarcoma in resource-limited settings: a three-arm, open-label, randomised, non-inferiority trial. Lancet. 2020 Apr 11;395(10231):1195-1207. doi: 10.1016/S0140-6736(19)33222-2. Epub 2020 Mar 5. PMID 32145827
- See also: DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 2.0, November 2014 — http://rsc.tech-res.com/docs/default-source/safety/daids_ae_grading_table_v2_nov2014.pdf?sfvrsn=8
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — http://rsc.tech-res.com/docs/default-source/safety/manual_for_expedited_reporting_aes_to_daids_v2.pdf?sfvrsn=12

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from October 2013 to March 2018 at 11 sites from Africa and South America (Brazil).
Groups:
- BV+ART: Bleomycin and Vincristine plus ART (co-formulated Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate)
- ET+ART: Etoposide plus ART (co-formulated Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate)
- PTX+ART: Paclitaxel plus ART (co-formulated Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate)
Period: Overall Study
Arm/Group | BV+ART | ET+ART | PTX+ART
Started | 135 | 60 | 139
Completed | 88 | 26 | 98
Not Completed | 47 | 34 | 41
Not completed — Death | 37 | 18 | 25
Not completed — Site is closing | 4 | 9 | 7
Not completed — Withdrew consent | 0 | 3 | 1
Not completed — Not willing to adhere to requirements | 0 | 2 | 3
Not completed — Not able to get to clinic | 2 | 0 | 2
Not completed — Severe debilitation, unable to continue | 0 | 0 | 1
Not completed — Unable to contact participant/parent | 1 | 1 | 1
Not completed — Enrollment Violation | 0 | 1 | 0
Not completed — Never started chemotherapy | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who were eligible for the study and who started their randomized chemotherapy.
Groups:
- Total: Total of all reporting groups
Arm/Group | BV+ART | ET+ART | PTX+ART | Total
Number analyzed (Participants) | 132 | 59 | 138 | 329
Age, Continuous [Median (Full Range); unit: years] | 35 [18 to 64] | 35 [23 to 72] | 35 [20 to 65] | 35 [18 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 14 | 31 | 76
  Male | 101 | 45 | 107 | 253
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7 | 14
  Not Hispanic or Latino | 127 | 57 | 131 | 315
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 130 | 58 | 136 | 324
  White | 2 | 1 | 2 | 5
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Malawi | 54 | 27 | 56 | 137
  Brazil | 5 | 2 | 7 | 14
  South Africa | 7 | 0 | 8 | 15
  Zimbabwe | 32 | 18 | 29 | 79
  Uganda | 7 | 10 | 9 | 26
  Kenya | 27 | 2 | 29 | 58
CD4 Cell Count, categorized [Count of Participants; unit: Participants] — CD4 cell count at screening.
  Participants
    <100 cells/mm^3 | 26 | 14 | 30 | 70
    >=100 cells/mm^3 | 106 | 45 | 108 | 259
Karnofsky Performance Score [Count of Participants; unit: Participants] — Karnofsky performance score at screening. Karnofsky performance score is from 0 (dead) to 100 (normal; no complaints; no evidence of disease) by increments of 10.
  Participants
    60 | 1 | 1 | 1 | 3
    70 | 11 | 7 | 14 | 32
    80 | 41 | 19 | 47 | 107
    90 | 79 | 32 | 75 | 186
    100 | 0 | 0 | 1 | 1
CD4 Cell Count [Median (Inter-Quartile Range); unit: cells/mm^3] — Mean of screening and entry CD4 cell count
  cells/mm^3 | 232 [134 to 369] | 216 [99 to 357] | 231 [127 to 341] | 229 [120 to 357]
HIV-1 RNA, continuous [Median (Inter-Quartile Range); unit: Log10 copies/mL] — HIV-1 RNA at entry
  Log10 copies/mL | 4.6 [2.7 to 5.2] | 4.9 [3.9 to 5.3] | 4.0 [2.5 to 5.1] | 4.4 [2.7 to 5.2]
HIV-1 RNA, categorized [Count of Participants; unit: Participants] — HIV-1 RNA at entry
  Participants
    <400 copies/mL | 29 | 4 | 38 | 71
    400 to <1,000 copies/mL | 14 | 2 | 10 | 26
    1000 to <10,000 copies/mL | 12 | 10 | 20 | 42
    >=10,000 copies/mL | 77 | 43 | 70 | 190
Number of Cutaneous KS Lesions [Count of Participants; unit: Participants] — At study entry
  Participants
    <=50 lesions | 32 | 21 | 51 | 104
    >50 lesions | 100 | 38 | 87 | 225
Presence of Oral Cavity KS Lesions [Count of Participants; unit: Participants] — At study entry
  Participants | 90 | 36 | 80 | 206
Presence of Lower Limb Edema [Count of Participants; unit: Participants] — At study entry
  Participants | 71 | 24 | 56 | 151
Presence of Lower Limb Edema in Both Limbs [Count of Participants; unit: Participants] — At study entry
  Participants | 39 | 11 | 22 | 72
Presence of Visceral KS [Count of Participants; unit: Participants] — At study entry
  Participants | 36 | 20 | 32 | 88

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Rate of Progression-Free Survival by Week 48 for ET+ART vs. PTX+ART
Description: Progression-free survival (PFS) by week 48 is defined as a lack of the following events: (a) Independent Endpoint Review Committee (IERC)-confirmed KS progression, (b) death, (c) entry into an additional step, or (d) loss to follow-up, prior to week 48. PFS rate was estimated by the Kaplan-Meier survival probability at week 48. Time to event was computed as the number of weeks from study entry to the first among these events. For participants who did not have any of the events, event time was censored at the week of last contact with the participant. Follow-up time beyond 48 was censored at week 48. Overall KS outcome status (complete response, partial response, stable, disease progression) was based on comparing follow-up to study entry or best KS response with respect to clinical assessment of KS cutaneous lesions (count, character and marker lesion area), oral KS, visceral KS and tumor-associated edema and as described in the publications (Krown et al 1989, Cianfrocca et al 2002).
Time Frame: From study entry to week 48
Population: All eligible participants who initiated study chemotherapy with available data as of March 2016.
Measure: Number (95% Confidence Interval); unit: Cumulative events per 100 persons
Arm/Group | ET+ART | PTX+ART
Number analyzed (Participants) | 59 | 59
Cumulative events per 100 persons | 19.7 [6.3 to 33.1] | 49.8 [32.4 to 67.3]
Statistical Analysis 1: Comparison: ET+ART vs PTX+ART; Treatment comparison was made using the difference (ET+ART - PTX+ART) in the stratified Kaplan-Meier estimate for the week 48 PFS rate with 95% two-sided confidence interval; Test type: Non-Inferiority — Non-inferiority is defined as demonstrating that the 48-week PFS rate in ET+ART is within 15 percent of PTX+ART. The selection of the 15 percent non-inferiority margin was a combination of clinical judgment and statistical reasoning. A poll of the sites was conducted to derive the "maximum treatment difference that is considered clinically relevant" (i.e. largest acceptable difference in order to gain the advantages (e.g. cost) of the experimental chemotherapy); Cumulative rate difference = -30.3, 95% CI 2-sided [-52.3 to -8.3] — Confidence interval (CI) estimation was stratified by screening CD4 count using Greenwood's variance with the inverse of this variance used for the stratum weights. CI stratified by country was not performed due to small number of observations

2. Primary Outcome: Cumulative Rate of Progression-Free Survival by Week 48 for BV+ART vs. PTX+ART
Description: as for outcome 1
Time Frame: From study entry to week 48
Population: All eligible participants who initiated study chemotherapy with available data as of March 2018.
Measure: Number (95% Confidence Interval); unit: Cumulative events per 100 persons
Arm/Group | BV+ART | PTX+ART
Number analyzed (Participants) | 132 | 138
Cumulative events per 100 persons | 44.1 [35.0 to 53.2] | 64.2 [55.4 to 73.0]
Statistical Analysis 1: Comparison: BV+ART vs PTX+ART; Treatment comparison was made using the difference (BV+ART - PTX+ART) in the stratified Kaplan-Meier estimate for the week 48 PFS rate with 95% two-sided confidence interval; Test type: Non-Inferiority — Non-inferiority is defined as demonstrating that the 48-week PFS rate in BV+ART is within 15 percent of PTX+ART. The selection of the 15 percent non-inferiority margin was a combination of clinical judgment and statistical reasoning. A poll of the sites was conducted to derive the "maximum treatment difference that is considered clinically irrelevant" (i.e. largest acceptable difference in order to gain the advantages (e.g. cost) of the experimental chemotherapy); Cumulative rate difference = -19.8, 95% CI 2-sided [-32.3 to -7.4] — Confidence interval estimation was stratified by screening CD4 count using Greenwood's variance with the inverse of this variance used for the stratum weights
Statistical Analysis 2: Comparison: BV+ART vs PTX+ART; Treatment comparison was made using the difference (BV+ART - PTX+ART) in the stratified Kaplan-Meier estimate for the week 48 cumulative PFS rate with 95% two-sided confidence interval; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Cumulative rate difference = -20.1, 95% CI 2-sided [-32.2 to -7.9] — Confidence interval estimation was stratified by country using Greenwood's variance with the inverse of this variance used for the stratum weights

3. Secondary Outcome: Cumulative Rate of Death by Week 48 for ET+ART vs. PTX+ART
Description: The Kaplan-Meier estimate of the cumulative rate of death by week 48. Time to death was computed as the number of weeks from study entry to date of death. For participants who did have the event, time to death was censored at the week of last contact with the participant. Time to death above 48 were censored at week 48.
Time Frame: From study entry to week 48
Population: All eligible participants who initiated study chemotherapy with available data as of March 2016.
Measure: Number (95% Confidence Interval); unit: Cumulative events per 100 persons
Arm/Group | ET+ART | PTX+ART
Number analyzed (Participants) | 59 | 59
Cumulative events per 100 persons | 25.6 [10.9 to 40.3] | 10.7 [2.6 to 18.8]
Statistical Analysis 1: Comparison: ET+ART vs PTX+ART; Treatment comparison was made using the difference (ET+ART - PTX+ART) in the stratified Kaplan-Meier estimate for the week 48 cumulative rate of death with 95% two-sided confidence interval; Test type: Other; Cumulative rate difference = 14.7, 95% CI 2-sided [-1.9 to 31.4] — Confidence interval estimation was stratified by screening CD4 lymphocyte count using Greenwood's variance with the inverse of this variance used for the stratum weights

4. Secondary Outcome: Cumulative Rate of Death by Week 48 for BV+ART vs. PTX+ART
Description: The Kaplan-Meier estimate of the cumulative rate of death by week 48. Time to death was computed as the number of weeks from study entry to the death date. For participants who did have the event, time to death was censored at the week of last contact with the participant. Time to death above 48 were censored at week 48.
Time Frame: From study entry to week 48
Population: All eligible participants who initiated study chemotherapy with available data as of March 2018.
Measure: Number (95% Confidence Interval); unit: Cumulative events per 100 persons
Arm/Group | BV+ART | PTX+ART
Number analyzed (Participants) | 132 | 138
Cumulative events per 100 persons | 18.5 [11.5 to 25.5] | 10.3 [5.0 to 15.7]
Statistical Analysis 1: Comparison: BV+ART vs PTX+ART; Treatment comparison was made using the difference (BV+ART - PTX+ART) in the stratified Kaplan-Meier estimate for the week 48 cumulative rate of death with 95% two-sided confidence interval; Test type: Other; Cumulative rate difference = 8.4, 95% CI 2-sided [-0.4 to 17.2] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Cumulative Rate of IERC-confirmed KS Progression by Week 48 for ET+ART vs. PTX+ART
Description: The Kaplan-Meier estimate of the cumulative rate of IERC-confirmed KS progression by week 48. IERC-confirmed KS progression was defined as KS disease progression confirmed by the IERC based on comparing follow-up KS response to study entry or best KS response with respect to clinical assessment of KS cutaneous lesions (count, character and marker lesion area), oral KS, visceral KS and tumor-associated edema and as described in the publications (Krown et al 1989, Cianfrocca et al 2002).
Time Frame: From study entry to week 48
Population: All eligible participants who initiated study chemotherapy with available data as of March 2016.
Measure: Number (95% Confidence Interval); unit: Cumulative events per 100 persons
Arm/Group | ET+ART | PTX+ART
Number analyzed (Participants) | 59 | 59
Cumulative events per 100 persons | 69.8 [54.2 to 85.3] | 41.2 [21.8 to 60.7]

6. Secondary Outcome: Cumulative Rate of IERC-confirmed KS Progression by Week 48 for BV+ART vs. PTX+ART
Description: as for outcome 5
Time Frame: From study entry to week 48
Population: All eligible participants who initiated study chemotherapy with available data as of March 2018.
Measure: Number (95% Confidence Interval); unit: Cumulative events per 100 persons
Arm/Group | BV+ART | PTX+ART
Number analyzed (Participants) | 132 | 138
Cumulative events per 100 persons | 43.9 [34.1 to 53.8] | 25.7 [17.1 to 34.3]
Statistical Analysis 1: Comparison: BV+ART vs PTX+ART; Treatment comparison was made using the difference (BV+ART - PTX+ART) in the stratified Kaplan-Meier estimate for the week 48 cumulative rate of IERC-confirmed KS progression with 95% two-sided confidence interval; Test type: Other; Cumulative rate difference = 16.3, 95% CI 2-sided [3.7 to 28.8]; Confidence interval estimation was stratified by screening CD4 lymphocyte count using Greenwood's variance with the inverse of this variance used for the stratum weights

7. Secondary Outcome: Cumulative Rate of AIDS-defining Event by Week 48 for ET+ART vs. PTX+ART
Description: The Kaplan-Meier estimate of the cumulative rate of AIDS-defining events by week 48. AIDS-defining events refer to non-KS AIDS-defining diagnosis (WHO Stage 4 (2007), plus microsporidiosis, cyclospora gastroenteritis, Chagas disease and visceral leishmaniasis). Time to event was computed as the number of weeks from study entry to the first AIDS-defining event. For participants who did not have any of the events, event time was censored at the week of last contact with the participant. Follow-up time beyond 48 was censored at week 48.
Time Frame: From study entry to week 48
Population: All eligible participants who initiated study chemotherapy with available data as of March 2016.
Measure: Number (95% Confidence Interval); unit: Cumulative events per 100 persons
Arm/Group | ET+ART | PTX+ART
Number analyzed (Participants) | 59 | 59
Cumulative events per 100 persons | 15.2 [3.8 to 26.6] | 28.6 [12.0 to 45.3]
Statistical Analysis 1: Comparison: ET+ART vs PTX+ART; Treatment comparison was made using the difference (ET+ART - PTX+ART) in the stratified Kaplan-Meier estimate for the week 48 cumulative rate of AIDS-defining events with 95% two-sided confidence interval; Test type: Other; Cumulative rate difference = -15.0, 95% CI 2-sided [-34.4 to 4.3] — [estimate comment as in outcome 3, analysis 1]

8. Secondary Outcome: Cumulative Rate of AIDS-defining Event by Week 48 for BV+ART vs. PTX+ART
Description: as for outcome 7
Time Frame: From study entry to week 48
Population: All eligible participants who initiated study chemotherapy with available data as of March 2018.
Measure: Number (95% Confidence Interval); unit: Cumulative events per 100 persons
Arm/Group | BV+ART | PTX+ART
Number analyzed (Participants) | 132 | 138
Cumulative events per 100 persons | 17.9 [10.7 to 25.1] | 19.6 [12.3 to 26.9]
Statistical Analysis 1: Comparison: BV+ART vs PTX+ART; Treatment comparison was made using the difference (BV+ART - PTX+ART) in the stratified Kaplan-Meier estimate for the week 48 cumulative rate of AIDS-defining events with 95% two-sided confidence interval; Test type: Other; Cumulative rate difference = -3.3, 95% CI 2-sided [-13.3 to 6.6] — [estimate comment as in outcome 3, analysis 1]

9. Secondary Outcome: Cumulative Rate of HIV-1 RNA Virologic Failure by Week 48 for ET+ART vs. PTX+ART
Description: Virologic failure is defined as two successive measurements of plasma HIV-1 RNA >=1000 copies/mL at week 12 to week 24 or RNA >=400 copies/mL at week 24 or later.
Time Frame: From study entry to week 48
Population: All eligible participants who initiated study chemotherapy with available data as of March 2016.
Measure: Number (95% Confidence Interval); unit: Cumulative events per 100 persons
Arm/Group | ET+ART | PTX+ART
Number analyzed (Participants) | 59 | 59
Cumulative events per 100 persons | 7.8 [0.0 to 16.4] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: ET+ART vs PTX+ART; Treatment comparison was made using the difference (ET+ART - PTX+ART) in the stratified Kaplan-Meier estimate for the week 48 cumulative rate of HIV-1 RNA virologic failure with 95% two-sided confidence interval; Test type: Other; Cumulative rate difference = 4.3, 95% CI 2-sided [-1.9 to 10.6] — [estimate comment as in outcome 3, analysis 1]

10. Secondary Outcome: Cumulative Rate of HIV-1 RNA Virologic Failure by Week 48 for BV+ART vs. PTX+ART
Description: as for outcome 9
Time Frame: From study entry to week 48
Population: All eligible participants who initiated study chemotherapy with available data as of March 2018.
Measure: Number (95% Confidence Interval); unit: Cumulative events per 100 persons
Arm/Group | BV+ART | PTX+ART
Number analyzed (Participants) | 132 | 138
Cumulative events per 100 persons | 7.4 [2.5 to 12.3] | 1.8 [0.0 to 4.2]
Statistical Analysis 1: Comparison: BV+ART vs PTX+ART; Treatment comparison was made using the difference (BV+ART - PTX+ART) in the stratified Kaplan-Meier estimate for the week 48 cumulative rate of HIV-1 RNA virologic failure with 95% two-sided confidence interval; Test type: Other; Cumulative rate difference = 5.5, 95% CI 2-sided [-0.1 to 11.0] — [estimate comment as in outcome 3, analysis 1]

11. Secondary Outcome: Number of Participants With Kaposi's Sarcoma-Immune Reconstitution Inflammatory Syndrome (KS-IRIS) for ET+ART vs. PTX+ART
Description: KS-IRIS is defined as any IERC-confirmed KS-progression that occurs within 12 weeks of ART-initiation that is associated with an increase in CD4 cell count of at least 50 cells/mm^3 above the study entry value and/or a decrease in the HIV-1 RNA level by at least 0.5 log below the study entry value prior to or at the time of documented KS progression.
Time Frame: From study entry to week 12
Population: All eligible participants who initiated study chemotherapy with available data as of March 2016.
Measure: Count of Participants; unit: Participants
Arm/Group | ET+ART | PTX+ART
Number analyzed (Participants) | 59 | 59
Participants | 6 | 0

12. Secondary Outcome: Number of Participants With Kaposi's Sarcoma-Immune Reconstitution Inflammatory Syndrome (KS-IRIS) for BV+ART vs. PTX+ART
Description: as for outcome 11
Time Frame: From study entry to week 12
Population: All eligible participants who initiated study chemotherapy with available data as of March 2018.
Measure: Count of Participants; unit: Participants
Arm/Group | BV+ART | PTX+ART
Number analyzed (Participants) | 132 | 138
Participants | 2 | 0

13. Secondary Outcome: Cumulative Rate of KS Progression, Death, or AIDS Defining Event by Week 48 for ET+ART vs. PTX+ART
Description: The Kaplan-Meier estimate of the cumulative rate of KS progression, death, or AIDS defining event by week 48
Time Frame: From study entry to week 48
Population: All eligible participants who initiated study chemotherapy with available data as of March 2016.
Measure: Number (95% Confidence Interval); unit: Cumulative events per 100 persons
Arm/Group | ET+ART | PTX+ART
Number analyzed (Participants) | 59 | 59
Cumulative events per 100 persons | 72.4 [58.1 to 86.8] | 54.6 [35.8 to 73.4]
Statistical Analysis 1: Comparison: ET+ART vs PTX+ART; Treatment comparison was made using the difference (ET+ART - PTX+ART) in the stratified Kaplan-Meier estimate for the week 48 cumulative rate of KS progression, death, or AIDS defining event; Test type: Other; Cumulative rate difference = 19.4, 95% CI 2-sided [-4.1 to 43.0] — [estimate comment as in outcome 3, analysis 1]

14. Secondary Outcome: Cumulative Rate of KS Progression, Death, or AIDS Defining Event by Week 48 for BV+ART vs. PTX+ART
Description: The Kaplan-Meier estimate of the cumulative rate of KS progression, death, or AIDS defining event by week 48
Time Frame: From study entry to week 48
Population: All eligible participants who initiated study chemotherapy with available data as of March 2018.
Measure: Number (95% Confidence Interval); unit: Cumulative events per 100 persons
Arm/Group | BV+ART | PTX+ART
Number analyzed (Participants) | 132 | 138
Cumulative events per 100 persons | 56.7 [47.6 to 65.7] | 42.1 [33.0 to 51.1]
Statistical Analysis 1: Comparison: BV+ART vs PTX+ART; Treatment comparison was made using the difference (BV+ART - PTX+ART) in the stratified Kaplan-Meier estimate for the week 48 cumulative rate of KS progression, death, or AIDS defining event; Test type: Other; Cumulative rate difference = 14.4, 95% CI 2-sided [1.8 to 27.0] — [estimate comment as in outcome 3, analysis 1]

15. Secondary Outcome: Cumulative Rate of KS Progression, Death, AIDS Defining Event, or Virologic Failure by Week 48 for ET+ART vs. PTX+ART
Description: The Kaplan-Meier estimate of the cumulative rate of KS progression, death, AIDS defining event, or virologic failure by week 48
Time Frame: From study entry to week 48
Population: All eligible participants who initiated study chemotherapy with available data as of March 2016.
Measure: Number (95% Confidence Interval); unit: Cumulative events per 100 persons
Arm/Group | ET+ART | PTX+ART
Number analyzed (Participants) | 59 | 59
Cumulative events per 100 persons | 77.5 [63.8 to 91.3] | 54.6 [35.8 to 73.4]
Statistical Analysis 1: Comparison: ET+ART vs PTX+ART; Treatment comparison was made using the difference (ET+ART - PTX+ART) in the stratified Kaplan-Meier estimate for the week 48 cumulative rate of KS progression, death, AIDS defining event, or virologic failure; Test type: Other; Cumulative rate difference = 24.2, 95% CI 2-sided [0.9 to 47.4] — [estimate comment as in outcome 3, analysis 1]

16. Secondary Outcome: Cumulative Rate of KS Progression, Death, AIDS Defining Event, or Virologic Failure by Week 48 for BV+ART vs. PTX+ART
Description: as for outcome 15
Time Frame: From study entry to week 48
Population: All eligible participants who initiated study chemotherapy with available data as of March 2018.
Measure: Number (95% Confidence Interval); unit: Cumulative events per 100 persons
Arm/Group | BV+ART | PTX+ART
Number analyzed (Participants) | 132 | 138
Cumulative events per 100 persons | 60.9 [51.9 to 69.8] | 42.0 [33.0 to 51.0]
Statistical Analysis 1: Comparison: BV+ART vs PTX+ART; Treatment comparison was made using the difference (BV+ART - PTX+ART) in the stratified Kaplan-Meier estimate for the week 48 cumulative rate of KS progression, death, AIDS defining event, or virologic failure; Test type: Other; Cumulative rate difference = 18.8, 95% CI 2-sided [6.3 to 31.3] — [estimate comment as in outcome 3, analysis 1]

17. Secondary Outcome: Cumulative Rate of KS Progression, Death, AIDS Defining Event, Virologic Failure, or KS-IRIS by Week 48 for ET+ART vs. PTX+ART
Description: The Kaplan-Meier estimate of the cumulative rate of KS progression, death, AIDS defining event, virologic failure, or KS-IRIS.
Time Frame: From study entry to week 48
Population: All eligible participants who initiated study chemotherapy with available data as of March 2016.
Measure: Number (95% Confidence Interval); unit: Cumulative events per 100 persons
Arm/Group | ET+ART | PTX+ART
Number analyzed (Participants) | 59 | 59
Cumulative events per 100 persons | 57.6 [45.0 to 70.2] | 33.9 [21.8 to 46.0]
Statistical Analysis 1: Comparison: ET+ART vs PTX+ART; Treatment comparison was made using the difference (ET+ART - PTX+ART) in the stratified Kaplan-Meier estimate for the week 48 cumulative rate of KS progression, death, AIDS defining event, virologic failure, or KS-IRIS; Test type: Other; Cumulative rate difference = 24.2, 95% CI 2-sided [0.9 to 47.4] — [estimate comment as in outcome 3, analysis 1]

18. Secondary Outcome: Cumulative Rate of KS Progression, Death, AIDS Defining Event, Virologic Failure, or KS-IRIS by Week 48 for BV+ART vs. PTX+ART
Description: as for outcome 17
Time Frame: From study entry to week 48
Population: All eligible participants who initiated study chemotherapy with available data as of March 2018.
Measure: Number (95% Confidence Interval); unit: Cumulative events per 100 persons
Arm/Group | BV+ART | PTX+ART
Number analyzed (Participants) | 132 | 138
Cumulative events per 100 persons | 54.5 [46.1 to 63.0] | 36.2 [28.2 to 44.3]
Statistical Analysis 1: Comparison: BV+ART vs PTX+ART; Treatment comparison was made using the difference (BV+ART - PTX+ART) in the stratified Kaplan-Meier estimate for the week 48 cumulative rate of KS progression, death, AIDS defining event, virologic failure, or KS-IRIS; Test type: Other; Cumulative rate difference = 17.7, 95% CI 2-sided [6.2 to 29.3] — [estimate comment as in outcome 3, analysis 1]

19. Secondary Outcome: Cumulative Rate of Change in KS Treatment by Week 48 for ET+ART vs. PTX+ART
Description: The Kaplan-Meier estimate of the cumulative rate of change in KS treatment by week 48. Change in KS treatment was defined as stopping Step 1 randomized chemotherapy and initiating a different chemotherapy.
Time Frame: From study entry to week 48
Population: All eligible participants who initiated study chemotherapy with available data as of March 2016.
Measure: Number (95% Confidence Interval); unit: Cumulative events per 100 persons
Arm/Group | ET+ART | PTX+ART
Number analyzed (Participants) | 59 | 59
Cumulative events per 100 persons | 59.5 [41.5 to 77.5] | 26.0 [8.8 to 43.3]
Statistical Analysis 1: Comparison: ET+ART vs PTX+ART; Treatment comparison was made using the difference (ET+ART - PTX+ART) in the stratified Kaplan-Meier estimate for the week 48 cumulative rate of change in KS treatment; Test type: Other; Cumulative rate difference = 37.5, 95% CI 2-sided [13.6 to 61.4] — [estimate comment as in outcome 3, analysis 1]

20. Secondary Outcome: Cumulative Rate of Change in KS Treatment by Week 48 for BV+ART vs. PTX+ART
Description: as for outcome 19
Time Frame: From study entry to week 48
Population: All eligible participants who initiated study chemotherapy with available data as of March 2018.
Measure: Number (95% Confidence Interval); unit: Cumulative events per 100 persons
Arm/Group | BV+ART | PTX+ART
Number analyzed (Participants) | 132 | 138
Cumulative events per 100 persons | 32.5 [23.3 to 41.7] | 18.9 [11.2 to 26.6]
Statistical Analysis 1: Comparison: BV+ART vs PTX+ART; Treatment comparison was made using the difference (BV+ART - PTX+ART) in the stratified Kaplan-Meier estimate for the week 48 cumulative rate of change in KS treatment; Test type: Other; Cumulative rate difference = 11.1, 95% CI 2-sided [-0.4 to 22.7] — [estimate comment as in outcome 3, analysis 1]

21. Secondary Outcome: Cumulative Rate of Death for ET+ART vs. PTX+ART
Description: The Kaplan-Meier estimate of the cumulative rate of death. Time to death was computed as the number of weeks between study entry and date of death. For participants who did not have the event, time to death was censored at the week of last contact with the participant or at the participant's off study week, whichever is later.
Time Frame: From study entry to week 240
Population: All eligible participants who initiated study chemotherapy with available data as of March 2016.
Measure: Number (95% Confidence Interval); unit: Cumulative events per 100 persons
Arm/Group | ET+ART | PTX+ART
Number analyzed (Participants) | 59 | 59
Cumulative events per 100 persons | 25.6 [10.9 to 40.3] | 10.7 [2.6 to 18.8]
Statistical Analysis 1: Comparison: ET+ART vs PTX+ART; Treatment comparison was made using the difference (ET+ART - PTX+ART) in the stratified Kaplan-Meier estimate for the cumulative rate of death with 95% two-sided confidence interval; Test type: Other; Cumulative rate difference = 14.7, 95% CI 2-sided [-1.9 to 31.4] — [estimate comment as in outcome 3, analysis 1]

22. Secondary Outcome: Cumulative Rate of Death for BV+ART vs PTX+ART
Description: as for outcome 21
Time Frame: From study entry to week 240
Population: All eligible participants who initiated study chemotherapy with available data as of March 2018.
Measure: Number (95% Confidence Interval); unit: Cumulative events per 100 persons
Arm/Group | BV+ART | PTX+ART
Number analyzed (Participants) | 132 | 138
Cumulative events per 100 persons | 18.5 [11.5 to 25.5] | 10.3 [5.0 to 15.7]
Statistical Analysis 1: Comparison: BV+ART vs PTX+ART; Treatment comparison was made using the difference (BV+ART - PTX+ART) in the stratified Kaplan-Meier estimate for the cumulative rate of death with 95% two-sided confidence interval; Test type: Other; Cumulative rate difference = 8.4, 95% CI 2-sided [-0.4 to 17.2] — [estimate comment as in outcome 3, analysis 1]

23. Secondary Outcome: Time to IERC-confirmed KS Progression or Death for ET+ART vs. PTX+ART
Description: Time to IERC-confirmed KS progression or death was computed as the number of weeks between study entry and the earlier between date of IERC-confirmed KS progression or date of death. For participants who did not have the event, event time was censored at the week of last contact with the participant or the participant's off study week, whichever is later. The 25-th percentile and hazard ratio are presented.
Time Frame: From study entry to week 240
Population: All eligible participants who initiated study chemotherapy with available data as of March 2016.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | ET+ART | PTX+ART
Number analyzed (Participants) | 59 | 59
weeks | 17.9 [8.9 to 22.0] | 30.0 [24.9 to 43.7]
Statistical Analysis 1: Comparison: ET+ART vs PTX+ART; Test type: Other; Hazard Ratio (HR) = 1.9, 95% CI 2-sided [1.1 to 3.4] — Hazard ratio for ET+ART relative to PTX+ART adjusted for screening CD4 lymphocyte count

24. Secondary Outcome: Time to IERC-confirmed KS Progression or Death for BV+ART vs. PTX+ART
Description: Time to IERC-confirmed KS progression or death was computed as the number of weeks between study entry and the earlier between date of IERC-confirmed KS progression or date of death. For participants who did not have the event, event time was censored at the week of last contact with the participant or at the participant's off study week, whichever is later.The 25-th percentile and hazard ratio are presented.
Time Frame: From study entry to week 240
Population: All eligible participants who initiated study chemotherapy with available data as of March 2018.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | BV+ART | PTX+ART
Number analyzed (Participants) | 132 | 138
weeks | 24.7 [21.3 to 30.0] | 38.6 [32.9 to 57.9]
Statistical Analysis 1: Comparison: BV+ART vs PTX+ART; Test type: Other; Hazard Ratio (HR) = 1.5, 95% CI 2-sided [1.1 to 2.2] — Hazard ratio for BV+ART relative to PTX+ART adjusted for screening CD4 lymphocyte count

25. Secondary Outcome: Number of Participants With Objective Response for ET+ART vs. PTX+ART
Description: The number of participants with objective response (complete response or partial response) as best overall KS response in Step 1. Overall KS response status (complete response, partial response, stable, disease progression) was based on comparing follow-up KS response to study entry or best KS response with respect to clinical assessment of KS cutaneous lesions (count, character and marker lesion area), oral KS, visceral KS and tumor-associated edema and as described in the publications (Krown et al 1989, Cianfrocca et al 2002).
Time Frame: From study entry up to week 144
Population: All eligible participants who initiated study chemotherapy with available data as of March 2016.
Measure: Count of Participants; unit: Participants
Arm/Group | ET+ART | PTX+ART
Number analyzed (Participants) | 59 | 59
Participants | 18 | 34
Statistical Analysis 1: Comparison: ET+ART vs PTX+ART; Test type: Other; Odds Ratio (OR) = 0.3, 95% CI 2-sided [0.1 to 0.7] — Odds ratio for ET+ART relative to PTX+ART adjusted for screening CD4 lymphocyte count

26. Secondary Outcome: Number of Participants With Objective Response for BV+ART vs. PTX+ART
Description: as for outcome 25
Time Frame: From study entry up to week 144
Population: All eligible participants who initiated study chemotherapy with available data as of March 2018.
Measure: Count of Participants; unit: Participants
Arm/Group | BV+ART | PTX+ART
Number analyzed (Participants) | 132 | 138
Participants | 80 | 91
Statistical Analysis 1: Comparison: BV+ART vs PTX+ART; Test type: Other; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.5 to 1.3] — Odds ratio for BV+ART relative to PTX+ART adjusted for screening CD4 lymphocyte count and country

27. Secondary Outcome: Duration of Objective Response for ET+ART vs. PTX+ART
Description: Duration of objective response is the number of weeks from first complete or partial response to the earliest among progression, death or off study week. The 25th percentile duration is presented.
Time Frame: From study entry up to week 144
Population: All eligible participants who initiated study chemotherapy with complete of partial KS response in Step 1 as of March 2016.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | ET+ART | PTX+ART
Number analyzed (Participants) | 18 | 34
weeks | 10.1 [3.0 to 24.0] | 19.9 [12.0 to 46.1]

28. Secondary Outcome: Duration of Objective Response for BV+ART vs. PTX+ART
Description: as for outcome 27
Time Frame: From study entry up to week 144
Population: All eligible participants who initiated study chemotherapy with complete of partial KS response in Step 1 as of March 2018.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | ET+ART | PTX+ART
Number analyzed (Participants) | 80 | 91
weeks | 21.0 [12.0 to 30.6] | 45.7 [22.4 to 56.7]

29. Secondary Outcome: Number of Participants With Symptomatic Peripheral Neuropathy (SPN)
Description: SPN consists of three assessments: (1) pain, aching or burning in feet, legs, (2) "pins and needles" in feet, legs, and (3) numbness (lack of feeling) in feet, legs. SPN is graded on a severity scale from 0 (not present), 1 (mild) to 10 (severe). Presence of SPN is defined as having grade >=1 in at least one of the three assessments.
Time Frame: Screening, Weeks 3, 6, 9, 12, 15, 18, 21. Assessment of SPN for ET+ART was only done at screening, weeks 9 and 21.
Population: All eligible participants who initiated study chemotherapy with available data as of March 2018.
Measure: Count of Participants; unit: Participants
Arm/Group | BV+ART | ET+ART | PTX+ART
Number analyzed (Participants) | 132 | 59 | 138
Participants
  Screening | 76 | 24 | 59
  Week 3: number analyzed (Participants) | 116 | 0 | 126
  Week 3 | 62 | 0 | 34
  Week 6: number analyzed (Participants) | 109 | 0 | 117
  Week 6 | 46 | 0 | 32
  Week 9: number analyzed (Participants) | 110 | 42 | 112
  Week 9 | 40 | 14 | 27
  Week 12: number analyzed (Participants) | 102 | 0 | 112
  Week 12 | 36 | 0 | 23
  Week 15: number analyzed (Participants) | 96 | 0 | 108
  Week 15 | 26 | 0 | 16
  Week 18: number analyzed (Participants) | 71 | 0 | 77
  Week 18 | 25 | 0 | 15
  Week 21: number analyzed (Participants) | 94 | 30 | 105
  Week 21 | 30 | 4 | 20

30. Secondary Outcome: Number of Participants With Peripheral Neuropathy (PN)
Description: Presence of PN is defined as having all of the following results: presence of symptomatic PN, abnormal perception of vibrations, and absent or hypoactive deep tendon reflexes.
Time Frame: Screening, Weeks 3, 6, 9, 12, 15, 18, 21. Assessment of PN for ET+ART was only done at screening, weeks 9 and 21.
Population: All eligible participants who initiated study chemotherapy with available data as of March 2018.
Measure: Count of Participants; unit: Participants
Arm/Group | BV+ART | ET+ART | PTX+ART
Number analyzed (Participants) | 132 | 59 | 138
Participants
  Screening | 7 | 1 | 0
  Week 3: number analyzed (Participants) | 116 | 0 | 126
  Week 3 | 1 | 0 | 0
  Week 6: number analyzed (Participants) | 109 | 0 | 117
  Week 6 | 1 | 0 | 2
  Week 9: number analyzed (Participants) | 110 | 42 | 112
  Week 9 | 3 | 0 | 2
  Week 12: number analyzed (Participants) | 102 | 0 | 112
  Week 12 | 3 | 0 | 4
  Week 15: number analyzed (Participants) | 96 | 0 | 108
  Week 15 | 2 | 0 | 3
  Week 18: number analyzed (Participants) | 71 | 0 | 77
  Week 18 | 6 | 0 | 1
  Week 21: number analyzed (Participants) | 94 | 30 | 105
  Week 21 | 5 | 0 | 2

31. Secondary Outcome: Number of Participants With Treatment-related Toxicities and Adverse Events (AEs)
Description: Adverse events classified by the site personnel as possibly, probably or definitely related to ART or chemotherapy.
Time Frame: From study entry to week 240
Population: All eligible participants who initiated study chemotherapy with available data as of March 2018.
Measure: Count of Participants; unit: Participants
Arm/Group | BV+ART | ET+ART | PTX+ART
Number analyzed (Participants) | 132 | 59 | 138
Participants
  Any Laboratory, Diagnosis or Signs/Symptoms | 32 | 25 | 48
  Any Laboratory | 27 | 25 | 39
  Any Diagnosis | 12 | 10 | 16
  Any Signs/Symptoms | 9 | 5 | 18

32. Secondary Outcome: Changes in CD4+ Lymphocyte Cell Count for ET+ART vs. PTX+ART
Description: Baseline CD4 lymphocyte cell count is the mean of screening and Step 1 entry CD4 values. Absolute change in CD4+ lymphocyte cell count was calculated as value at a given visit minus the baseline CD4 lymphocyte cell count.
Time Frame: Baseline, weeks 12, 24, 48
Population: All eligible participants who initiated study chemotherapy with available data as of March 2016.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | ET+ART | PTX+ART
Number analyzed (Participants) | 59 | 59
cells/mm^3
  Week 12 CD4 change: number analyzed (Participants) | 38 | 43
  Week 12 CD4 change | 37 [-4 to 83] | 47 [12 to 97]
  Week 24 CD4 change: number analyzed (Participants) | 24 | 32
  Week 24 CD4 change | 106 [-4 to 136] | 95 [24 to 179]
  Week 48 CD4 change: number analyzed (Participants) | 5 | 12
  Week 48 CD4 change | 69 [19 to 122] | 157 [25 to 338]

33. Secondary Outcome: Changes in CD4+ Lymphocyte Cell Count for BV+ART vs. PTX+ART
Description: as for outcome 32
Time Frame: Baseline, weeks 12, 24, 48
Population: All eligible participants who initiated study chemotherapy with available data as of March 2018.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | BV+ART | PTX+ART
Number analyzed (Participants) | 132 | 138
cells/mm^3
  Week 12 CD4 change: number analyzed (Participants) | 108 | 114
  Week 12 CD4 change | 21 [-43 to 70] | 37 [-6 to 97]
  Week 24 CD4 change: number analyzed (Participants) | 95 | 103
  Week 24 CD4 change | 43 [-25 to 110] | 65 [-1 to 159]
  Week 48 CD4 change: number analyzed (Participants) | 46 | 66
  Week 48 CD4 change | 112 [11 to 172] | 105 [21 to 177]

34. Secondary Outcome: Self-reported Adherence to ART Therapy
Description: ART adherence is based on participant's recall of the number of missed ART doses for the past month. Perfect adherence is defined as having zero missed ART doses.
Time Frame: At Weeks 6, 12, 18, 30 and 48
Population: All eligible participants who initiated study chemotherapy with available data as of March 2018.
Measure: Count of Participants; unit: Participants
Arm/Group | BV+ART | ET+ART | PTX+ART
Number analyzed (Participants) | 132 | 59 | 138
Participants
  Week 6 Perfect Adherence: number analyzed (Participants) | 114 | 49 | 122
  Week 6 Perfect Adherence | 101 | 43 | 106
  Week 12 Perfect Adherence: number analyzed (Participants) | 108 | 38 | 112
  Week 12 Perfect Adherence | 101 | 36 | 103
  Week 18 Perfect adherence: number analyzed (Participants) | 98 | 35 | 110
  Week 18 Perfect adherence | 85 | 29 | 97
  Week 30 Perfect adherence: number analyzed (Participants) | 73 | 16 | 94
  Week 30 Perfect adherence | 66 | 13 | 85
  Week 48 Perfect adherence: number analyzed (Participants) | 17 | 0 | 21
  Week 48 Perfect adherence | 13 | 0 | 20

35. Secondary Outcome: Presence of Oral KS
Description: Funding for oral KS objectives including data and sample collection was withdrawn during the study conduct.
Time Frame: From study entry to week 240
Population: The corresponding outcome measure was withdrawn.
Arm/Group | BV+ART | ET+ART | PTX+ART
Number analyzed (Participants) | 0 | 0 | 0

36. Secondary Outcome: Salivary KSHV
Description: Funding for oral KS objectives including data and sample collection was withdrawn during the study conduct.
Time Frame: Baseline, weeks 60, 120, 180, 240
Population: The corresponding outcome measure was withdrawn.
Arm/Group | BV+ART | ET+ART | PTX+ART
Number analyzed (Participants) | 0 | 0 | 0

37. Secondary Outcome: Number of Participants With IERC-Confirmed KS Disease Progression, Dose-Limiting Toxicity, Death, AIDS-Defining Events, Virologic Failure and Objective Response in Step 2
Description: IERC-confirmed KS progression refers to KS disease progression confirmed by the IERC based on comparing follow-up KS response to study entry or best KS response with respect to clinical assessment of KS cutaneous lesions (count, character and marker lesion area), oral KS, visceral KS and tumor-associated edema and as described in the publications (Krown et al 1989, Cianfrocca et al 2002). AIDS-defining events refer to non-KS AIDS-defining diagnosis (WHO Stage 4 (2007), plus microsporidiosis, cyclospora gastroenteritis, Chagas disease and visceral leishmaniasis). Virologic failure is defined as two successive measurements of plasma HIV-1 RNA >=1000 copies/mL at week 12 to week 24 or RNA >=400 copies/mL at week 24 or later. Objective response refers to complete response or partial response as best overall KS response. Results are presented by Step 2 treatment arm.
Time Frame: From Step 2 study entry to Step 2 discontinuation, up to 144 weeks
Population: All eligible participants who entered Step 2 with available data as of March 2018.
Measure: Count of Participants; unit: Participants
Arm/Group | BV+ART | ET+ART | PTX+ART
Number analyzed (Participants) | 10 | 1 | 9
Participants
  With IERC-confirmed KS progression | 1 | 1 | 1
  With dose-limiting toxicity | 0 | 0 | 0
  Died | 1 | 0 | 5
  With AIDS-defining events | 1 | 0 | 0
  With virologic failure | 2 | 1 | 1
  With objective response | 7 | 0 | 5

38. Secondary Outcome: Number of Participants With IERC-Confirmed KS Disease Progression, Dose-Limiting Toxicity, Death, AIDS-Defining Events, Virologic Failure and Objective Response in Step 3
Description: IERC-confirmed KS progression refers to KS disease progression confirmed by the IERC based on comparing follow-up KS response to study entry or best KS response with respect to clinical assessment of KS cutaneous lesions (count, character and marker lesion area), oral KS, visceral KS and tumor-associated edema and as described in the publications (Krown et al 1989, Cianfrocca et al 2002). AIDS-defining events refer to non-KS AIDS-defining diagnosis (WHO Stage 4 (2007), plus microsporidiosis, cyclospora gastroenteritis, Chagas disease and visceral leishmaniasis). Virologic failure is defined as two successive measurements of plasma HIV-1 RNA >=1000 copies/mL at week 12 to week 24 or RNA >=400 copies/mL at week 24 or later. Objective response refers to complete response or partial response as best overall KS response. Results are presented by Step 3 treatment arm.
Time Frame: From Step 3 study entry to Step 3 discontinuation, up to 144 weeks
Population: All eligible participants who entered Step 3 with available data as of March 2018.
Measure: Count of Participants; unit: Participants
Arm/Group | BV+ART | ET+ART | PTX+ART
Number analyzed (Participants) | 29 | 6 | 42
Participants
  With IERC-confirmed KS progression | 6 | 2 | 8
  With dose-limiting toxicity | 0 | 0 | 0
  Died | 3 | 0 | 7
  With AIDS-defining events | 5 | 0 | 7
  With virologic failure | 2 | 2 | 1
  With objective response | 18 | 5 | 29

39. Secondary Outcome: Number of Participants With IERC-Confirmed KS Disease Progression, Dose-Limiting Toxicity, Death, AIDS-Defining Events, Virologic Failure and Objective Response in Step 4
Description: IERC-confirmed KS progression refers to KS disease progression confirmed by the IERC based on comparing follow-up KS response to study entry or best KS response with respect to clinical assessment of KS cutaneous lesions (count, character and marker lesion area), oral KS, visceral KS and tumor-associated edema and as described in the publications (Krown et al 1989, Cianfrocca et al 2002). AIDS-defining events refer to non-KS AIDS-defining diagnosis (WHO Stage 4 (2007), plus microsporidiosis, cyclospora gastroenteritis, Chagas disease and visceral leishmaniasis). Virologic failure is defined as two successive measurements of plasma HIV-1 RNA >=1000 copies/mL at week 12 to week 24 or RNA >=400 copies/mL at week 24 or later. Objective response refers to complete response or partial response as best overall KS response. Results are presented by Step 4 treatment arm.
Time Frame: From Step 4 study entry to Step 4 discontinuation, up to 96 weeks
Population: All eligible participants who entered Step 4 with available data as of March 2018.
Measure: Count of Participants; unit: Participants
Arm/Group | BV+ART | PTX+ART
Number analyzed (Participants) | 5 | 6
Participants
  With IERC-confirmed KS progression | 2 | 3
  With dose-limiting toxicity | 0 | 0
  Died | 3 | 2
  With AIDS-defining events | 0 | 0
  With virologic failure | 1 | 0
  With objective response | 3 | 3

40. Other Pre Specified Outcome: Quality of Life Measures
Description: The protocol did not distinguish between outcome measures essential to the primary publication and those of lesser importance and priority which are not the focus of the study but intended for subsequent publications of exploratory analyses, conditional on primary results and additional funding. This outcome measure was listed under secondary outcome measures in the study protocol but was intended for an exploratory analysis to compare measures of quality of life in ET+ART, BV+ART and PTX+ART.
Time Frame: Baseline, weeks 60, 120, 180, 240
Reporting Status: Not Posted

41. Other Pre Specified Outcome: Immunohistochemical Evaluations of Viral and Cellular Gene Expression
Description: The protocol did not distinguish between outcome measures essential to the primary publication and those of lesser importance and priority which are not the focus of the study but intended for subsequent publications of exploratory analyses, conditional on primary results and additional funding. This outcome measure was listed under secondary outcome measures in the study protocol but was intended for an exploratory analysis to evaluate the relationship between response of KS to therapy and development of KS-IRIS with immunohistochemical markers of viral and cellular gene expression in KS tumors. The laboratory assays for this outcome measure have not been completed.
Time Frame: Baseline, 24-48 hours after 2nd chemo-therapy cycle begins
Reporting Status: Not Posted

42. Other Pre Specified Outcome: RNA Levels for KSHV Genes
Description: The protocol did not distinguish between outcome measures essential to the primary publication and those of lesser importance and priority which are not the focus of the study but intended for subsequent publications of exploratory analyses, conditional on primary results and additional funding. This outcome measure was listed under secondary outcome measures in the study protocol but was intended for an exploratory analysis to evaluate the relationship between response of KS to therapy and development of KS-IRIS with RNA levels for KSHV genes in tumor biopsies. The laboratory assays for this outcome measure have not been completed.
Time Frame: Baseline, weeks 60, 120, 180, 240
Reporting Status: Not Posted

43. Other Pre Specified Outcome: Cellular and Humoral Markers of Immune Function and Activation
Description: The protocol did not distinguish between outcome measures essential to the primary publication and those of lesser importance and priority which are not the focus of the study but intended for subsequent publications of exploratory analyses, conditional on primary results and additional funding. This outcome measure was listed under secondary outcome measures in the study protocol but was intended for an exploratory analysis to evaluate the relationship between response of KS to therapy and development of KS-IRIS with cellular and humoral markers of immune function and activation. The laboratory assays for this outcome measure have not been completed.
Time Frame: Baseline, weeks 60, 120, 180, 240
Reporting Status: Not Posted

44. Other Pre Specified Outcome: Plasma KS-associated Herpesvirus (KSHV)
Description: The protocol did not distinguish between outcome measures essential to the primary publication and those of lesser importance and priority which are not the focus of the study but intended for subsequent publications of exploratory analyses, conditional on primary results and additional funding. This outcome measure was listed under secondary outcome measures in the study protocol but was intended for an exploratory analysis to investigate the relationship between plasma and PBMC KSHV viral load. The laboratory assays for this outcome measure have not been completed.
Time Frame: Baseline, weeks 60, 120, 180, 240
Reporting Status: Not Posted

45. Other Pre Specified Outcome: Peripheral Blood Mononuclear Cell (PBMC) KSHV
Description: as for outcome 44
Time Frame: Baseline, weeks 60, 120, 180, 240
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From study entry to off study date, average follow-up time of 96 weeks, maximum of 209 weeks.
Description: The study protocol required reporting of all new diagnoses, signs/symptoms >=Grade 3, lab toxicities >=Grade 2, and all signs/symptoms and lab toxicities that led to a change in treatment, regardless of grade. All signs/symptoms, lab results, or diagnostic test results observed or performed as part of establishing a diagnosis were requested regardless of grade. The DAIDS AE Grading Table (V1.0) and EAE Manual (V2.0) were used. All eligible participants who initiated study treatment are included.
Groups:
- Bleomycin Plus Vincristine (BV) Plus Co-formulated EFV/FTC/TDF: Bleomycin and Vincristine plus ART (co-formulated Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate)
- Etoposide (ET) Plus Co-formulated EFV/FTC/TDF: Etoposide plus ART (co-formulated Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate)
- Paclitaxel (PTX) Plus Co-formulated EFV/FTC/TDF: Paclitaxel plus ART (co-formulated Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate)
Arm/Group | Bleomycin Plus Vincristine (BV) Plus Co-formulated EFV/FTC/TDF | Etoposide (ET) Plus Co-formulated EFV/FTC/TDF | Paclitaxel (PTX) Plus Co-formulated EFV/FTC/TDF
All-Cause Mortality (participants affected / at risk) | 37/132 | 33/59 | 55/138
Serious Adverse Events (participants affected / at risk) | 54/132 | 33/59 | 55/138
Other Adverse Events (participants affected / at risk) | 130/132 | 58/59 | 133/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bleomycin Plus Vincristine (BV) Plus Co-formulated EFV/FTC/TDF (N=132) | Etoposide (ET) Plus Co-formulated EFV/FTC/TDF (N=59) | Paclitaxel (PTX) Plus Co-formulated EFV/FTC/TDF (N=138)
Anaemia (Blood and lymphatic system disorders) | 9 | 2 | 8
Bicytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 6 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Death (General disorders) | 7 | 2 | 5
Drowning (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 6 | 4 | 6
Cellulitis (Infections and infestations) | 2 | 1 | 0
Central nervous system infection (Infections and infestations) | 0 | 0 | 1
Chronic hepatitis B (Infections and infestations) | 0 | 1 | 0
Disseminated tuberculosis (Infections and infestations) | 0 | 1 | 1
Encephalitis (Infections and infestations) | 0 | 1 | 0
Extrapulmonary tuberculosis (Infections and infestations) | 0 | 2 | 0
Gangrene (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 2
HIV infection WHO clinical stage IV (Infections and infestations) | 0 | 0 | 1
Immune reconstitution inflammatory syndrome associated tuberculosis (Infections and infestations) | 1 | 1 | 0
Malaria (Infections and infestations) | 1 | 1 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0
Meningitis cryptococcal (Infections and infestations) | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 2 | 6
Pneumonia bacterial (Infections and infestations) | 4 | 2 | 3
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 1 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 3
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 2 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Transaminases increased (Investigations) | 1 | 0 | 1
Weight decreased (Investigations) | 1 | 1 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 10 | 9
Facial paralysis (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 0
Abortion complete (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bleomycin Plus Vincristine (BV) Plus Co-formulated EFV/FTC/TDF (N=132) | Etoposide (ET) Plus Co-formulated EFV/FTC/TDF (N=59) | Paclitaxel (PTX) Plus Co-formulated EFV/FTC/TDF (N=138)
Anaemia (Blood and lymphatic system disorders) | 5 | 6 | 3
Abdominal pain (Gastrointestinal disorders) | 5 | 5 | 9
Diarrhoea (Gastrointestinal disorders) | 9 | 8 | 17
Gastritis (Gastrointestinal disorders) | 3 | 3 | 1
Vomiting (Gastrointestinal disorders) | 13 | 9 | 13
Asthenia (General disorders) | 7 | 2 | 4
Chest pain (General disorders) | 13 | 5 | 13
Malaise (General disorders) | 3 | 3 | 4
Mucosal discolouration (General disorders) | 9 | 4 | 1
Oedema peripheral (General disorders) | 17 | 3 | 13
Pain (General disorders) | 13 | 5 | 6
Peripheral swelling (General disorders) | 6 | 5 | 5
Pyrexia (General disorders) | 26 | 14 | 22
Bacterial sepsis (Infections and infestations) | 12 | 5 | 5
Gastroenteritis (Infections and infestations) | 2 | 4 | 1
Malaria (Infections and infestations) | 7 | 2 | 5
Pneumonia bacterial (Infections and infestations) | 10 | 3 | 13
Pulmonary tuberculosis (Infections and infestations) | 7 | 4 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 6 | 7
Urinary tract infection (Infections and infestations) | 5 | 5 | 3
Alanine aminotransferase increased (Investigations) | 14 | 5 | 16
Aspartate aminotransferase increased (Investigations) | 20 | 15 | 29
Blood albumin decreased (Investigations) | 84 | 40 | 86
Blood alkaline phosphatase increased (Investigations) | 23 | 9 | 23
Blood bicarbonate decreased (Investigations) | 21 | 9 | 22
Blood bilirubin increased (Investigations) | 7 | 4 | 5
Blood creatinine increased (Investigations) | 14 | 9 | 13
Blood glucose decreased (Investigations) | 8 | 4 | 6
Blood glucose increased (Investigations) | 20 | 11 | 24
Blood phosphorus decreased (Investigations) | 18 | 9 | 26
Blood potassium increased (Investigations) | 5 | 3 | 1
Blood sodium decreased (Investigations) | 58 | 31 | 62
Carbon dioxide decreased (Investigations) | 8 | 9 | 3
Haemoglobin decreased (Investigations) | 47 | 29 | 48
Neutrophil count decreased (Investigations) | 42 | 29 | 55
Platelet count decreased (Investigations) | 27 | 10 | 21
Weight decreased (Investigations) | 23 | 10 | 17
White blood cell count decreased (Investigations) | 6 | 6 | 13
Decreased appetite (Metabolism and nutrition disorders) | 11 | 4 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 | 11 | 17
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 8 | 11
Headache (Nervous system disorders) | 14 | 7 | 6
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 7
Acute kidney injury (Renal and urinary disorders) | 1 | 5 | 3
Dysuria (Renal and urinary disorders) | 5 | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 13 | 27
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 8 | 10
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 7
Skin ulcer (Skin and subcutaneous tissue disorders) | 5 | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT01435018/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/18/NCT01435018/SAP_001.pdf